CLINICAL TRIAL: NCT03228836
Title: Efficacy and Safety Evaluation of IBI308 in Patients With Relapsed/Refractory Extranodal NK/T Cell Lymphoma, Nasal Type: a Multicenter, Single Arm, Phase 2 Study (ORIENT-4)
Brief Title: Efficacy and Safety Evaluation of IBI308 in Patients With Extranodal NK/T Cell Lymphoma Patients
Acronym: ORIENT-4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI308D201
Record Dates: First submitted 2017-07-22; First posted 2017-07-25 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Effect of Drugs
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab (IBI308) (Experimental)
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Sintilimab (IBI308) 200mg IV Q3W

SUMMARY:
This is phase II study. Efficacy and safety evaluation of IBI308 in patients with relapsed/refractory extranodal NK/T cell lymphoma, nasal type: a multicenter, single arm.

DETAILED DESCRIPTION:
Extranodal NK/T cell lymphoma, nasal type(ENKTL) accounts for about 6% of all lymphomas in china. Epstein Barr virus (EBV) infection is found in all cases of ENKTL and maybe plays an important pathogenetic role.

Conventional anthrocycline-based regimens are not preferred to be used in ENKTL because of high p-glycoprotein expression. ORR of L-asparaginase based regimens is about 80% and no salvage regimens are recommended in ENKTL so far after failure of L-asparaginase based regimen.

Recently, a phase II clinical trial result demonstrated high ORR of anti-PD-1 antibody treatment in ENKTL.IBI308, a humanized monoclonal antibody (mAb) directly against PD-1, is investigated in this phase II Chinese ENKTL clinical trial.

Additionally the correlation between PD-L1 expression and the response to IBI308 treatment in Chinese ENKTL subjects will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

1. Histologically confirmed ENKL-NT.
2. Relapsed or refractory ENKTL-NT. Being relapsed is defined as presence of new lesions at the primary location or other sites after achieving CR; being refractory is defined as any one of the followings: PD after 2 treatment cycles, PR not achieved after 4 treatment cycles, or CR not achieved after 6 treatment cycles. Patients who do not response or patients with relapsed disease or PD after autologous stem cell transplantation can enroll.
3. Must have been treated with asparaginase-based regimen (radiotherapy must be performed for stage I/II disease).
4. Long axis of a lesion > 15 mm or 18FDG-PET uptake by lesion.
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) scores of 0-2.
6. Signed the inform consent form (ICF) and able to comply with the scheduled follow-up visits and related procedures required in the protocol.
7. Between the ages of ≥18 to ≤70 years.
8. Life expectancy≥ 12 weeks.
9. Patients (female patients at childbearing age or male patients whose partners are at childbearing age) must take effective contraceptive measures during the entire course of the trial and within 90 days since the last dose of treatment.
10. Adequate organs and bone marrow functions, as defined below: Count of whole blood cells: absolute neutrophil count (ANC) ≥1.0×10^9/L, platelets (PLTs) count ≥ 50×10^9/L, hemoglobin (HGB) ≥ 8.0 g/L; granulocyte colony-stimulating factor, PLT, or red blood cell (RBC) transfusion has not been performed within 7 days prior to the test. Hepatic function: total bilirubin (TBIL) ≤ 1.5×upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN. Renal function:serum creatinine (Cr) ≤ 1.5 × ULN. Thyroid function: normal thyroid stimulating hormone (TSH) at baseline, or abnormal TSH at baseline with normal thiiodothronine (T3)/thiiodothronine (T4) and no symptoms.

Exclusion Criteria:

1. Patients with aggressive NK cell leukemia.
2. Patients with primary or secondary central nervous system (CNS) lymphoma.
3. Patients with severe hemophagocytic syndrome at initial diagnosis of ENKTL-NT.
4. Patients with pulmonary great vessel invasion.
5. Previous exposure to any anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies.
6. Enrolled in another interventional clinical study, unless only involved in an observational study (non-interventional) or in the follow-up phase of an interventional study.
7. Received any investigational drug within 4 weeks prior to the first dose of study treatment.
8. The last dose of radiation or anti-tumor therapy (chemotherapy, targeted therapy or tumor embolization) was within 3 weeks prior to receiving the first dose of study treatment; the last dose of nitrosourea or mitomycin C treatment was within 6 weeks prior to receiving the first dose of study treatment.
9. Received immunosuppressants within 4 weeks prior to the first dose of study treatment, excluding local glucocorticoids administered by nasal, inhaled, or other topical routes, or systemic glucocorticoids of physiological doses (no more than 10 mg/day of prednisone or equivalents).
10. Received any live attenuated vaccine within 4 weeks prior to the first dose of study treatment, or is scheduled to receive live attenuated vaccine during the study period.
11. Received major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study treatment, or has unhealed wounds, ulcers, or fractures.
12. Active, known, or suspected autoimmune disease (see Appendix 6) or previous medical history of these diseases within 2 years (patients with vitiligo, psoriasis, alopecia, or Graves' disease not requiring systemic treatment, hypothyroidism only requiring thyroid replacement, or type I diabetes only requiring insulin can enroll).
13. Known history of primary immunodeficiency diseases.
14. Known active pulmonary tuberculosis.
15. Known history of allogeneic organ transplantation or allogeneic hem atopoietic stem cell transplantation.
16. Known to be allergic to any ingredients of monoclonal antibodies.
17. Uncontrolled concurrent diseases including but not limited to:

    HIV-infected patients (positive anti-HIV antibody). Active or poorly controlled severe infections. Symptomatic congestive heart failure (NYHA Class III-IV) or symptomatic or poorly controlled arrhythmia.

    Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg) despite of standard treatment.

    Any arterial thromboembolic events occurred within 6 months prior to enrollment, including myocardial infarction, unstable angina, cerebrovascular accident, or transient cerebral ischemic attack.

    Life-threatening hemorrhagic events or grade 3-4 gastrointestinal/variceal hemorrhage requiring blood transfusion, endoscopy, or surgical treatment within 3 months prior to enrollment.

    History of deep venous thrombosis, pulmonary embolism, or other serious thromboembolic events within 3 months prior to enrollment (implantable port or catheter-related thrombosis, or superficial venous thrombosis are not considered as serious thromboembolisms).

    Uncontrolled metabolic disorders, non-malignant organ or systemic diseases, or cancer-related secondary diseases that may lead to higher medical risks and/or survival evaluation uncertainties.

    Hepatic encephalopathy, hepatorenal syndrome, or cirrhosis with Child-Pugh grade B or C.

    Bowel obstruction or history of the following diseases: inflammatory bowel disease or extensive bowel resection (partial colectomy or extensive small bowel resection accompanied with chronic diarrhea), Crohn's disease, and ulcerative colitis.

    Acute or chronic diseases, psychiatric disorders, or laboratory abnormalities that may lead to the following consequences: increased investigational drug-related risks, or interference with interpreting trial results, and considered ineligible for participating in the trial by the investigators.
18. Known acute or chronic active hepatitis B (chronic HBV carriers or inactive HBsAg-positive patients can enroll if the HBV DNA < 1×10^3 copies/mL), or acute or chronic active hepatitis C (patients with negative HCV antibody can enroll; HCV RNA test is required for patients with positive HCV antibody, those test negative can enroll).
19. History of GI perforation and/or fistula without radical treatment within 6 months prior to the enrollment.
20. Known interstitial lung disease.
21. Clinically uncontrollable third spacing, such as pleural effusion and ascites that cannot be controlled by drainage or other methods prior to enrollment.
22. History of other primary malignant tumors, excluding:

    History of radical treatment for malignant tumors with no evidence of tumor recurrence for more than 5 years prior to enrollment and with a very low risk of recurrence.

    Adequately treated nonmelanoma skin cancer or lentigo maligna with no signs of disease recurrence.

    Adequately treated carcinoma in situ with no signs of disease recurrence.
23. Pregnant or breastfeeding female patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian-yong Li, Master, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Provincial Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tao R, Fan L, Song Y, Hu Y, Zhang W, Wang Y, Xu W, Li J. Sintilimab for relapsed/refractory extranodal NK/T cell lymphoma: a multicenter, single-arm, phase 2 trial (ORIENT-4). Signal Transduct Target Ther. 2021 Oct 27;6(1):365. doi: 10.1038/s41392-021-00768-0. PMID 34702811

RESULTS

PARTICIPANT FLOW:
Groups:
- Sintilimab (IBI308): Participants with relapsed or refractory ENKTL-NT were enrolled to receive sintilimab (IBI308) 200mg intravenous infusion (IV) every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | Sintilimab (IBI308)
Started | 28
Treated | 28
Completed | 11
Not Completed | 17
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Disease Progression | 7
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Groups:
- Sintilimab (IBI308): Participants with relapsed or refractory ENKTL-NT were enrolled to receive sintilimab (IBI308) 200mg IV Q3W.
Arm/Group | Sintilimab (IBI308)
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.32 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 28
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 28

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Before First PD
Description: The tumor assessment is according to Lugano 2014 Criteria and then International Working Group (IWG) 2007 Criteria after 24 weeks. Objective response is defined as best overall response (CR or PR) across all assessment time points during the period from enrollment to termination of trial treatment (per Lugano 2014 criteria during intial 24 weeks, per IWG 2007 criteria after 24 weeks). The primary efficacy endpoint is ORR evaluated using the 2014 Lugano Criteria before first progression disease (PD).
Time Frame: Up to ~30 months (through database cut-off date of 28-February-2020)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sintilimab (IBI308)
Number analyzed (Participants) | 28
Percentage of Participants | 60.7 [40.6 to 78.5]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the first dose to the first documented progressive disease (PD) per Lugano 2014 or death due to any cause, whichever occurred first. Participates who neither progress nor die were censored at the date of their last tumor imaging evaluation. Participates who did not have any tumor imaging evaluation after baseline were censored on the date of enrollment.
Time Frame: Up to ~30 months (through database cut-off date of 28-February-2020)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sintilimab (IBI308)
Number analyzed (Participants) | 28
Days | 104.0 [45.0 to 419.0]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from first date of response to first PD per Lugano 2014 or death. Subjects who neither progress nor die were censored at the date of their last tumor imaging evaluation.
Time Frame: Up to ~30 months (through database cut-off date of 28-February-2020)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sintilimab (IBI308)
Number analyzed (Participants) | 28
Days | 126.0 [64.0 to 463.0]

ADVERSE EVENTS:
Time Frame: Up to ~30 months (through database cut-off date of 28-February-2020)
Description: Safety Population: all the participants who received at least one dose of the investigational drug.
Groups:
- Sintilimab (IBI308): Sintilimab (IBI308) 200mg IV Q3W
Arm/Group | Sintilimab (IBI308)
All-Cause Mortality (participants affected / at risk) | 7/28
Serious Adverse Events (participants affected / at risk) | 7/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sintilimab (IBI308) (N=28)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
Pyrexia (General disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Localised infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sintilimab (IBI308) (N=28)
Anaemia (Blood and lymphatic system disorders) | 3
Lymphadenitis (Blood and lymphatic system disorders) | 2
Myocardial ischaemia (Cardiac disorders) | 2
Ventricular extrasystoles (Cardiac disorders) | 3
Autoimmune thyroiditis (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 9
Constipation (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 2
Face oedema (General disorders) | 2
Pain (General disorders) | 2
Pyrexia (General disorders) | 13
Enterovirus infection (Infections and infestations) | 2
Gingivitis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 5
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 5
Blood albumin decreased (Investigations) | 5
Blood alkaline phosphatase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 5
Blood glucose increased (Investigations) | 7
Blood lactate dehydrogenase increased (Investigations) | 6
Blood thyroid stimulating hormone increased (Investigations) | 8
C-reactive protein increased (Investigations) | 2
Electrocardiogram abnormal (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 2
Globulins decreased (Investigations) | 2
Globulins increased (Investigations) | 5
Haemoglobin decreased (Investigations) | 9
Haemoglobin urine present (Investigations) | 2
Lipase increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 17
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 6
Protein total decreased (Investigations) | 2
Protein urine present (Investigations) | 4
Red blood cells urine positive (Investigations) | 2
Thyroid function test abnormal (Investigations) | 2
Thyroxine free decreased (Investigations) | 5
Thyroxine increased (Investigations) | 4
Tri-iodothyronine free decreased (Investigations) | 2
Urine ketone body present (Investigations) | 2
Weight decreased (Investigations) | 2
White blood cell count decreased (Investigations) | 14
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT03228836/Prot_001.pdf
  • Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT03228836/SAP_002.pdf